CLINICAL TRIAL: NCT02810587
Title: Incidence of Endophthalmitis After Intravitreous Anti-vascular Endothelial Growth Factor Injections Comparison Between Patients Receiving Versus Not Receiving Topical Antibiotics Following the Injections
Brief Title: Endophthalmitis After Intravitreous Anti-VEGF Injections in Patients Receiving vs. Not Receiving Topical Antibiotics
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Voraporn Chaikitmongkol, Instructor, Chiang Mai University
Other Study IDs: OPT-2558-02789
Record Dates: First submitted 2016-06-16; First posted 2016-06-23 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-06

CONDITIONS: Endophthalmitis
Keywords: Endophthalmitis; Intravitreous injection; anti-vascular endothelial growth factor; topical antibiotics
MeSH Terms: conditions — Endophthalmitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Topical antibiotics group: Those who receive topical antibiotics after intravitreous injection as home medication for 7 days.
  Interventions: Drug: Topical antibiotics following injection
- No topical antibiotics group: Those who does NOT receive topical antibiotics after intravitreous injection as home medication.

INTERVENTIONS:
Drug: Topical antibiotics following injection — Either receive or not receive topical antibiotics following intravitreous injection
  Groups: Topical antibiotics group

SUMMARY:
This is a prospective case series which aims to determine the incidence of endophthalmitis following intravitreous anti-vascular endothelial growth factor (VEGF) injection comparing between eyes receiving post-injection antibiotics drops and those not receiving antibiotics drops treated at Chiang Mai University Hospital between May 2015 and April 2017 (2-year period).

DETAILED DESCRIPTION:
Intravitreous anti-VEGF injection has been the most common procedure performed at eye clinics worldwide. It becomes the gold standard treatment for many macular diseases, such as diabetic macular edema and neovascular age-related macular degeneration (AMD). One of the most serious complication after intravitreous injection is post-injection endophthalmitis. There is no proven preventive strategy of post-injection endophthalmitis except the use of povidone iodine. However, a number of physicians around the world prescribe topical antibiotics after the injection, despite the lack of evidence to support the benefit of topical antibiotics to prevent the occurence of endophthalmitis. Recently, many large trials from the US including the Diabetic Retinopathy Clinical Research Network (DRCR.net), the Comparison of AMD Treatment Trials (CATT) study have reported the incidence of post-injection endophthalmitis comparing between eyes receiving versus not receiving post-injection antibiotics, and the results of all studies suggested that topical antibiotics does not help reduce the incidence of post-injection endophthalmitis. In addition, the results suggested that eyes receiving antibiotics had higher rate of endophthalmitis comparing to those not receiving antibiotics. Therefore, a majority of physicians in the United States have stopped prescribing antibiotics drops following the injection. However, a majority of physicians in Asia-Pacific region still prescribe antibiotics drops following the injection (according to the Preferences and Trends (PAT) survey by the American Society of Retina Specialists in 2014).

Due to the limited evidence from Asian literature whether there is difference between incidence of endophthalmitis following intravitreous anti-VEGF injection between eyes receiving antibiotics drops versus not receiving antibiotics drops in the Asian setting, the investigators conducted this study to determine the incidence of endophthalmitis after intravitreous anti-VEGF injection, comparing between eyes receiving post-injection antibiotics versus not receiving. Results from this study would be beneficial to guide an appropriate practice for physicians in the Asian region.

ELIGIBILITY:
Inclusion Criteria:

1. More than 18 years of age
2. Have an eye conditions requiring intravitreous anti-VEGF injections, including neovascular age-related macular degeneration, diabetic macular edema, macular edema due to retinal vein occlusions in one or both eyes
3. Able to revisit for an eye evaluation at a recommended period (at least 3 weeks following the injection)
4. No history of uveitis or endophthalmitis in the study eye

Exclusion Criteria:

* Presence of blepharitis or conjunctivitis in the study at the time of intravitreous injection

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All of patients receiving intravitreous anti-vascular endothelial growth factors injections at Department of Ophthalmology, Faculty of Medicine, Chiang Mai University, between May 2015 and April 2017, who give consent and agree to follow up within the recommended period
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2015-05; Primary Completion 2017-04 (Estimated); Study Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of endophthalmitis | at least 3 weeks after the injection
  Endophthalmitis is defined as a presence of severe inflammation in the anterior chamber and vitreous cavity, associated with pain, redness, or any degree of decreased vision.

CONTACTS AND LOCATIONS:
Locations (1):
- Voraporn Chaikitmongkol, Muang Chiang Mai, Chiang Mai, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Storey P, Dollin M, Pitcher J, Reddy S, Vojtko J, Vander J, Hsu J, Garg SJ; Post-Injection Endophthalmitis Study Team. The role of topical antibiotic prophylaxis to prevent endophthalmitis after intravitreal injection. Ophthalmology. 2014 Jan;121(1):283-289. doi: 10.1016/j.ophtha.2013.08.037. Epub 2013 Oct 18. PMID 24144453
- [Result] Bhatt SS, Stepien KE, Joshi K. Prophylactic antibiotic use after intravitreal injection: effect on endophthalmitis rate. Retina. 2011 Nov;31(10):2032-6. doi: 10.1097/IAE.0b013e31820f4b4f. PMID 21659941
- [Result] Cheung CS, Wong AW, Lui A, Kertes PJ, Devenyi RG, Lam WC. Incidence of endophthalmitis and use of antibiotic prophylaxis after intravitreal injections. Ophthalmology. 2012 Aug;119(8):1609-14. doi: 10.1016/j.ophtha.2012.02.014. Epub 2012 Apr 4. PMID 22480743
- [Result] Bhavsar AR, Stockdale CR, Ferris FL 3rd, Brucker AJ, Bressler NM, Glassman AR; Diabetic Retinopathy Clinical Research Network. Update on risk of endophthalmitis after intravitreal drug injections and potential impact of elimination of topical antibiotics. Arch Ophthalmol. 2012 Jun;130(6):809-10. doi: 10.1001/archophthalmol.2012.227. No abstract available. PMID 22801859
- [Result] Bhavsar AR, Googe JM Jr, Stockdale CR, Bressler NM, Brucker AJ, Elman MJ, Glassman AR; Diabetic Retinopathy Clinical Research Network. Risk of endophthalmitis after intravitreal drug injection when topical antibiotics are not required: the diabetic retinopathy clinical research network laser-ranibizumab-triamcinolone clinical trials. Arch Ophthalmol. 2009 Dec;127(12):1581-3. doi: 10.1001/archophthalmol.2009.304. PMID 20008710